CLINICAL TRIAL: NCT00899496
Title: Pilot Study of Cancer Resistance in Humans
Brief Title: Laboratory Assay in Determining Cancer Resistance in Patients With Metastatic Cancer and in Healthy Participants
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU 95A05; P30CA012197 (NIH); CCCWFU-99A05; CCCWFU-BG05-342
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: stage IV bladder cancer; stage IV colon cancer; stage IV non-small cell lung cancer; stage IV pancreatic cancer; stage IV rectal cancer; stage IV renal cell cancer; stage IV melanoma; stage III multiple myeloma; extensive stage small cell lung cancer; stage IV adult soft tissue sarcoma; stage III malignant testicular germ cell tumor; stage IV breast cancer; stage IV ovarian epithelial cancer; stage IV prostate cancer; stage IV endometrial carcinoma; unspecified adult solid tumor, protocol specific; metastatic osteosarcoma; stage IV uterine sarcoma; stage III ovarian epithelial cancer; ovarian sarcoma; stage IV adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; cutaneous B-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; adult grade III lymphomatoid granulomatosis; primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Melanoma; Multiple Myeloma; Sarcoma; Testicular Neoplasms; Breast Neoplasms; Carcinoma, Ovarian Epithelial; Prostatic Neoplasms; Endometrial Neoplasms; Osteosarcoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Intraocular Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: immunological diagnostic method
Other: physiologic testing

SUMMARY:
RATIONALE: Studying samples of blood and tissue in the laboratory from patients with cancer and from healthy participants may help doctors learn more about cancer.

PURPOSE: This laboratory study is looking at an assay in determining cancer resistance in patients with metastatic cancer and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Optimize and standardize the in vitro cell kill assay using human white blood cells and human cancer cell lines from patients with metastatic cancer and from healthy participants.
* Determine the results of the in vitro cell kill assay in patients with metastatic cancer and in healthy participants with no history of cancer.

OUTLINE: This is a pilot study.

Peripheral blood is obtained from healthy participants and from cancer patients. Tissue is collected from archived samples. White blood cells are obtained from tissue and blood samples and are assessed by the in vitro cell kill assay.

PROJECTED ACCRUAL: A total of 24 patients and 24 healthy participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

-Meets 1 of the following criteria:

* Diagnosis of metastatic cancer including, but not limited to, any of the following:

  * Stage IV non-small cell lung cancer
  * Extensive-stage small cell lung cancer
  * Metastatic testicular cancer
  * Stage IV breast carcinoma
  * Stage III or IV ovarian carcinoma
  * Stage IV endometrial carcinoma
  * Stage IV prostate carcinoma
  * Stage IV colorectal or pancreatic cancer
  * Stage IV renal cancer
  * Stage III or IV non-Hodgkin's lymphoma
  * Stage IV bladder cancer
  * Stage III multiple myeloma (Salmon-Durie staging)
  * Metastatic melanoma
  * Metastatic sarcoma
* Healthy participant, meeting the following criteria:

  * No prior cancer
  * Over 50 years of age

Exclusion Criteria:

* Serious medical or psychiatric condition that would preclude study compliance
* Chemotherapy or radiotherapy within the past 3 months (patient)
* Prior immunosuppressive therapy or radiotherapy for any disease (healthy participant)

Max Age: 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those with metastatic cancer OR healthy individuals with no prior cancer diagnosis and who are over the age of 50.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2009-10-23 (Actual); Study Completion 2009-10-23 (Actual)

PRIMARY OUTCOMES:
Cell killing ability (positive or negative) | Day 180
Percentage of cells killed | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Cui, PhD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States